CLINICAL TRIAL: NCT01525238
Title: A Randomized, Multi-Center, Parallel Group, Single-Dose, Pharmacokinetics and Pharmacodynamics Study of Dapagliflozin in Children and Adolescents Aged 10 to 17 Years With Type 2 Diabetes Mellitus
Brief Title: PK Study of Dapagliflozin in Pediatric Subjects With T2DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MB102-091; 2011-005225-40 (EudraCT Number)
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dapagliflozin 2.5 mg (Experimental)
  Interventions: Drug: Dapagliflozin
- Dapagliflozin 5 mg (Experimental)
  Interventions: Drug: Dapagliflozin
- Dapagliflozin 10 mg (Experimental)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Tablet, Oral, 2.5 mg, Single-dose
  Arms: Dapagliflozin 2.5 mg
Drug: Dapagliflozin — Tablet, Oral, 5 mg, Single-dose
  Arms: Dapagliflozin 5 mg
Drug: Dapagliflozin — Tablet, Oral, 10 mg, Single-dose
  Arms: Dapagliflozin 10 mg

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics (PK) of Dapagliflozin in pediatric subjects with type 2 diabetes mellitus (T2DM)

DETAILED DESCRIPTION:
Primary purpose: The primary purpose is to assess the pharmacokinetics of a single dose of Dapagliflozin in the range of 2.5 to 10 mg in pediatric subjects aged 10 to 17 years with T2DM

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2DM
* Male and female subjects ages 10-17
* Glycosylated Hemoglobin A1c (HbA1c) ≥6 to 10%
* Body weight ≥30 kg

Exclusion Criteria:

* Fasting plasma glucose (FPG) >240 mg/dL at screening
* Abnormal renal function
* Active liver disease and/or significant abnormal liver function

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2014-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (14):
  - The Children Hospital Of Alabama, Birmingham, Alabama
  - Axis Clinical Trials, Los Angeles, California
  - Nemours Childrens Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Lsuhsc-Shreveport, Shreveport, Louisiana
  - Childrens Mercy Hospital, Kansas City, Missouri
  - Women And Children'S Hopsital Of Buffalo, Buffalo, New York
  - Promedica Toledo Children'S Hospital, Toledo, Ohio
  - Mercy Children'S Hospital, Toledo, Ohio
  - Children'S Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Children'S Hospital Of Pittsburgh Of Upmc, Pittsburgh, Pennsylvania
  - Methodist Le Bonheur Hlthcare, Memphis, Tennessee
  - Christus Santa Rosa Childrens Hospital, San Antonio, Texas
- Mexico (3):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Veracruz

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 53 participants enrolled; 24 randomized; 24 treated with study drug. 29 participants were not randomized due to no longer meeting study criteria (25), withdrawal of consent (2), or other reasons (2).
Period: Overall Study
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Started | 8 | 8 | 8
Completed | 7 | 8 | 8
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.69) | 14.0 (2.39) | 14.6 (2.13) | 14.5 (2.04)
Age, Customized [Number; unit: participants]
  10 to <= 15 years | 5 | 5 | 4 | 14
  16 to <= 17 years | 3 | 3 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 15
  Male | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean of Maximum Observed Plasma Concentration (Cmax) of Dapagliflozin
Description: Maximum observed plasma concentration (Cmax) was measured by plasma concentration of Dapagliflozin over time. The geometric means are reported in nanograms per milliliter (ng/mL).
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable pharmacokinetic (PK) profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
ng/mL | 24.8 (34) | 48.4 (41) | 118 (35)

2. Primary Outcome: Median Time of Maximum Observed Plasma Concentration (Tmax) of Dapagliflozin
Description: Time of maximum observed plasma concentration (Tmax) for Dapagliflozin was derived from plasma concentrations versus time data. Medians were reported in hours (h).
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles.
Measure: Median (Full Range); unit: hours
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
hours | 1.50 [0.75 to 2.00] | 0.960 [0.58 to 1.53] | 0.875 [0.75 to 4.00]

3. Primary Outcome: Geometric Mean of Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time [AUC(INF)] of Dapagliflozin
Description: Area under the plasma concentration-time curve from time zero extrapolated to infinite time was derived from concentration versus time data. Geometric means are reported in nanogram hours per milliliter (ng*hr/mL).
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
ng*h/mL | 101 (23) | 199 (29) | 427 (31)

4. Primary Outcome: Geometric Mean of Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-T)] of Dapagliflozin
Description: Area under the concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) was measured by plasma concentration of Dapagliflozin over time. The geometric means are reported in nanogram hours per milliliter (ng*h/mL).
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
ng*h/mL | 92.3 (27) | 189 (31) | 418 (31)

5. Primary Outcome: Mean Plasma Half-life (T-HALF) of Dapagliflozin
Description: Plasma half-life (T-Half) for Dapagliflozin was derived from plasma concentrations versus time data. Means are reported in hours.
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
hours | 14.1 (5.59) | 10.3 (3.72) | 10.7 (2.16)

6. Primary Outcome: Geometric Mean of Apparent Clearance After Extravascular Administration (CL/F) of Dapagliflozin
Description: Apparent clearance after extravascular administration (CL/F) of Dapagliflozin was derived from plasma concentrations versus time data. Geometric means are reported in milliliters per minute (mL/min).
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
mL/min | 413 (26) | 418 (27) | 391 (25)

7. Primary Outcome: Geometric Mean of Apparent Volume of Distribution at Terminal Phase After Extravascular Administration (Vz/F) of Dapagliflozin
Description: Geometric mean of apparent volume of distribution at terminal phase after extravascular administration of Dapagliflozin was derived from plasma concentration versus time data. Geometric means are reported in Liters (L)
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
Liters | 468 (34) | 343 (45) | 355 (34)

8. Secondary Outcome: Geometric Mean of Maximum Observed Plasma Concentration (Cmax) of Dapagliflozin 3-O-Glucuronide
Description: Maximum observed plasma concentration (Cmax) was measured by plasma concentration of Dapagliflozin 3-O-Glucuronide over time. The geometric means are reported in nanograms per milliliter (ng/mL).
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
ng/mL | 24.6 (45) | 49.0 (50) | 154 (27)

9. Secondary Outcome: Median Time of Maximum Observed Plasma Concentration (Tmax) of Dapagliflozin 3-O-Glucuronide
Description: Time of maximum observed plasma concentration (Tmax) for Dapagliflozin 3-O-Glucuronide was derived from plasma concentrations versus time data. Medians were reported in hours (h).
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Median (Full Range); unit: hours
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
hours | 1.50 [1.00 to 4.00] | 1.50 [0.83 to 4.00] | 1.50 [1.47 to 4.00]

10. Secondary Outcome: Geometric Mean of Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time [AUC(INF)] of Dapagliflozin 3-O-Glucuronide
Description: as for outcome 3
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
ng*hr/mL | 105 (23) | 232 (30) | 658 (21)

11. Secondary Outcome: Geometric Mean of Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-T)] of Dapagliflozin 3-O-Glucuronide
Description: Area under the concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) was measured by plasma concentration of Dapagliflozin 3-O-Glucuronide over time. The geometric means are reported in nanogram hours per milliliter (ng*h/mL).
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
ng*h/mL | 95.8 (20) | 208 (32) | 612 (24)

12. Secondary Outcome: Mean Plasma Half-life (T-HALF) of Dapagliflozin 3-O-Glucuronide
Description: Plasma half-life (T-Half) for Dapagliflozin was derived from plasma concentration versus time data. Means are reported in hours.
Time Frame: 11 time points: Immediately pre-dose, 0.5, 0.75, 1.0, 1.5, 4, 8, 12, 14, 24, and 48 hours post-dose
Population: All treated participants with evaluable PK profiles
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 7 | 8 | 8
hours | 4.62 (3.086) | 8.71 (2.024) | 8.37 (3.330)

13. Secondary Outcome: Mean Fasting Plasma Glucose Concentrations at Pre-dose on Day 1 and on Day 2 After an 8-hr Fasting
Description: Plasma glucose concentrations were evaluated in all treated subjects at Day 1 pre-dose and at Day 2 after fasting for 8 hours. Means are reported in milligrams per deciliter (mg/dL).
Time Frame: Day 1 (Pre-dose) to Day 2
Population: All treated participants with evaluable pharmacodynamic (PD) profiles
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 6 | 8 | 8
mg/dL
  Day 1 Pre-dose (n= 6, 8, 8) | 146.2 (72.56) | 152.1 (49.06) | 139.8 (39.63)
  Day 2 after 8 hour fast (n= 3, 8, 7) | 124.0 (45.21) | 119.4 (17.18) | 119.0 (29.15)

14. Secondary Outcome: Mean Change in Fasting Plasma Glucose From Baseline Until Day 2
Description: Plasma glucose concentrations were evaluated in all treated subjects at Day 1 pre-dose and at Day 2 after fasting for 8 hours. Mean change from baseline to Day 2 is reported in milligrams per deciliter (mg/dL).
Time Frame: Day 1 (Pre-dose) to Day 2
Population: All treated participants with evaluable PD profiles
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 3 | 8 | 7
mg/dL | -46.7 (60.08) | -32.8 (42.41) | -22.0 (27.32)

15. Secondary Outcome: Mean Total Amount of Glucose Excreted in Urine Over 24 Hours
Description: The total amount of glucose excreted in urine was measured for 24 hours following administration of Dapagliflozin. Means are reported in grams.
Time Frame: Time of dose to 24 hours post-dose, Day 1 to Day 2
Population: All treated participants with evaluable PD profiles
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 5 | 8 | 7
grams | 52.84 (27.18) | 62.39 (26.55) | 89.04 (41.25)

16. Secondary Outcome: Number of Participants With Vital Sign Abnormalities, Electrocardiogram (ECG) Abnormalities, or Physical Examination Abnormalities Following Study Drug Administration.
Description: Participants were followed from dosing on Day 1 until study discharge on Day 3. The number of participants with investigator-assessed clinically-important abnormalities in vital sign measurements, ECGs or physical examinations was reported.
Time Frame: Day 1 to Day 3
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 8 | 8 | 8
participants
  Vital sign abnormalities | 0 | 0 | 0
  ECG abnormalities | 0 | 0 | 0
  Physical examination abnormalities | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Marked Hematology Laboratory Abnormalities
Description: LLN=Lower Limit of Normal, ULN=Upper Limit of Normal, Pre-Rx=Value before first dose (Day -1). Lab values that met the following criteria were marked as abnormalities: Hemoglobin (grams per deciliter:g/dL): <0.85*Pre-Rx. Hematocrit (%): <0.85*Pre-Rx. Platelet Count (x10^9 cells per liter:c/L): <0.85*LLN or >1.5*ULN (if Pre-Rx<LLN, use <0.85*Pre-Rx). Leukocytes (x10^3 cells per microliter: c/uL): <0.9*LLN, >1.2*ULN (if Pre-Rx<LLN, use <0.85*Pre-Rx or >ULN, if Pre- Rx>ULN, use >1.15*Pre-Rx or <LLN). Neutrophils (Absolute) (x10^3 c/uL): <=1.5. Lymphocytes (Absolute) (x10^3 c/uL): <0.75 or >7.5. Monocytes (Absolute) (x10^3 c/uL): >2.000. Basophils (x10^3 c/uL): >0.4. Eosinophils (Absolute) (x10^3 c/uL): >0.75. Blasts (Absolute) (x10^9 c/L) > 0.
Time Frame: Day 1 (Pre-dose) to Day 3
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 8 | 8 | 8
participants
  Leukocytes, low (n=8, 8, 8) | 1 | 0 | 1
  Neutrophils, low (n=8, 8, 8) | 0 | 0 | 1

18. Secondary Outcome: Number of Participants With Marked Serum Chemistry Abnormalities
Description: LLN=Lower Limit of Normal, ULN=Upper Limit of Normal, Pre-Rx=Value before first dose. Lab values that met the following criteria were marked as abnormalities: Alkaline Phosphatase (units per liter: U/L), Aspartate Aminotransferase (U/L), Alanine Aminotransferase (U/L): >1.25*ULN (if Pre-Rx>ULN, use >1.25*Pre-Rx). Bilirubin (milligrams per deciliter: mg/dL): >1.1*ULN (if Pre-Rx>ULN, use >1.25*Pre-Rx). Blood Urea Nitrogen (mg/dL): >1.1*ULN (if Pre-Rx>ULN, use >1.2*Pre-Rx). Creatinine (micromoles per Liter (umol/L)): >1.5*ULN if Pre-Rx missing or <= ULN, >1.33*Pre-Rx if PreRx > ULN. Sodium (mmol/L): >1.05*ULN, 1.05*Pre-Rx if Pre-Rx>ULN: <0.95*Pre-Rx, >ULN. If Pre-Rx>ULN: >1.05*Pre-Rx, <LLN). Potassium(mmol/L), Chloride (mmol/L), Calcium(mmol/L): <0.9*LLN, >1.1*ULN (if Pre-Rx<LLN: <0.9*Pre-Rx, >ULN. If Pre-Rx>ULN: >1.1*Pre-Rx, <LLN). Phosphorus (mg/dL): <0.85*LLN, >1.25*ULN (if Pre-Rx<LLN, <0.85*Pre-Rx, >ULN. if Pre-Rx>ULN: >1.25*Pre-Rx, <LLN).
Time Frame: Day 1 (Pre-dose) to Day 3
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 8 | 8 | 8
participants
  ALT, high (8, 8, 8) | 1 | 0 | 0
  AST, high (n=8, 8, 8) | 1 | 0 | 0

19. Secondary Outcome: Number of Participants With Marked Abnormalities in Other Chemistry Testing
Description: LLN=Lower Limit of Normal, ULN=Upper Limit of Normal, Pre-Rx=Value before first dose. Lab values that met the following criteria were marked as abnormalities: Glucose, fasting serum (mmol/L): <0.8*LLN, >1.3*ULN (if Pre-Rx<LLN: <0.8*Pre-Rx, >ULN. If Pre-Rx>ULN: >2.0*Pre-Rx, <LLN). Protein (grams per deciliter: g/L): <0.9*LLN, >1.1*ULN (if Pre-Rx<LLN: <0.9*Pre-Rx, >ULN. If Pre-Rx>ULN: >1.1*Pre-Rx, <LLN). Albumin (g/L): <0.9*LLN (if Pre-Rx<LLN: <0.9*Pre-Rx). Uric Acid (mmol/L): >1.2*ULN (if Pre-Rx>ULN: >1.25*Pre-Rx). Lactate Dehydrogenase (U/L): >1.25*ULN (if Pre-Rx>ULN: >1.5*Pre-Rx)
Time Frame: Day 1 (Pre-dose) to Day 3
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 8 | 8 | 8
participants
  Glucose, fasting serum, high (n=7, 7, 7) | 1 | 1 | 0
  Additional other chemistry marked abnormalities | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Marked Urinalysis Abnormalities
Description: LLN=Lower Limit of Normal, ULN=Upper Limit of Normal, Pre-Rx=Value before first dose. Lab values that met the following criteria were marked as abnormalities: Blood, urine (Qualitative): >=2 (If Pre-Rx >= 1, >=2*Pre-Rx). Glucose, urine (Qualitative): >=1, (If Pre-Rx >=1, >=2*Pre-Rx). Protein, urine (Qualitative): >=2 (If Pre-Rx >=1, >=2*Pre-Rx). Red Blood Cells (RBC), urine (RBC per High Power Field (hpf)): >=2 (If Pre-Rx>=2, >=4). White Blood Cells (WBC), urine (hpf): >=2 (If Pre-Rx>=2, >=4).
Time Frame: Day 1 (Pre-dose) to Day 3
Population: All treated participants with evaluable lab results
Measure: Number; unit: participants
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 8 | 8 | 8
participants
  Blood, urine, high (n=8, 8, 8) | 0 | 0 | 2
  Glucose, urine, high (n=8, 8, 8) | 2 | 3 | 4
  Protein, urine, high (n=8, 8, 8) | 0 | 0 | 3
  RBC, urine, high (n=1, 1, 4) | 0 | 0 | 3
  WBC, urine, high (n=4, 2, 3) | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: SAEs collected from Screening (up to 28 days before first dose) to 30 days after last dose; Non-serious AEs collected from time of dose (Day 1) to Study Discharge (Day 3) and followed until resolution, stabilization, or reclassification as SAE.
Arm/Group | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 2.5 mg (N=8) | Dapagliflozin 5 mg (N=8) | Dapagliflozin 10 mg (N=8)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No